CLINICAL TRIAL: NCT00431691
Title: Effect of Antioxidants on Ocular Blood Flow, Endothelial Function, and Cytokine Levels in LPS Induced Inflammatory Model in Humans.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Wolzt, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-110106
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Retina; Regional Blood Flow; Endotoxin, Escherichia Coli
MeSH Terms: conditions — Escherichia coli Infections | interventions — Vitamins; endotoxin, Escherichia coli; Lipopolysaccharides; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: vitamin and mineral supplement; Drug: Escherichia coli Endotoxin (LPS); Drug: 100% O2; Drug: nitroglycerin
- 2 (Placebo Comparator)
  Interventions: Drug: Escherichia coli Endotoxin (LPS); Drug: 100% O2; Drug: nitroglycerin

INTERVENTIONS:
Drug: vitamin and mineral supplement — dose: 4 tablets daily for two weeks
  vitamin A 7160 IU, vitamin C 113mg, vitamin E 100IU, zinc 17.4mg, copper 0.4mg
  Other Names: Ocuvite preservision
  Arms: 1
Drug: Escherichia coli Endotoxin (LPS) — dose: 2 ng/kg (corresponding to 20 IU/kg), intravenous bolus over 5 minutes on both study days
  Other Names: US Standard Endotoxin
Drug: 100% O2 — breathing for 30 minutes, 2 breathing periods on both study days
Drug: nitroglycerin — dose: 0,8 mg sublingual, applied during FMD measurements on both study days
  Other Names: Nitrolingual Pump Spray

SUMMARY:
Oxidative stress, which refers to cellular damage caused by reactive oxygen intermediates, has been implicated in many disease processes, especially age-related disorders. Many trials investigating use of antioxidants in protecting different tissues against oxidative stress have been conducted, but the results are ambiguous.

Inflammation is generally associated with enhanced oxidative stress and widespread endothelial dysfunction. In the present study, the infusion of LPS, which is a cell wall component of Gram-negative bacteria and a major mediator in the pathogenesis of septic shock, will be used as a standardized experimental model of systemic inflammatory response in humans. The assessment of outcome parameters will include measurements of ocular blood flow, forearm blood flow and plasma concentration of cytokines. Measurements of ocular hemodynamics provide an unique chance to investigate local blood flow in humans non-invasively. Moreover, the retina is especially susceptible to oxidative stress because of its high consumption of oxygen, its high polyunsaturated fatty acid content, and its exposure to visible light. Evidence from literature clearly supports a role for oxidative stress in pathophysiology of several ocular diseases including diabetic retinopathy and age-related macular degeneration. To investigate the retinal vascular reactivity we will use systemic hyperoxia as a stimulus. The measurement of forearm blood flow will be use to assess endothelial function. The main study objective is to investigate the effect of oral vitamins and minerals supplementation on impaired retinal vascular reactivity after LPS administration.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug, vitamins and minerals supplements as well
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Retinal blood flow | in total 8x on 2 study days

SECONDARY OUTCOMES:
Choroidal blood flow | in total 4x on 2 study days
Flow mediated dilation (FMD) of brachial artery assessed with ultrasound | in total 4x on 2 study days
Blood pressure, heart rate | on 2 study days
Body temperature | on 2 study days
Concentration of cytokines in plasma | on 2 study days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pemp B, Polska E, Karl K, Lasta M, Minichmayr A, Garhofer G, Wolzt M, Schmetterer L. Effects of antioxidants (AREDS medication) on ocular blood flow and endothelial function in an endotoxin-induced model of oxidative stress in humans. Invest Ophthalmol Vis Sci. 2010 Jan;51(1):2-6. doi: 10.1167/iovs.09-3888. Epub 2009 Aug 13. PMID 19684008